CLINICAL TRIAL: NCT07112560
Title: Early Detection and Prevention of Amblyopia and Visual Impairment Through Systematic Pediatric Vision Screening
Acronym: FALSSE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9746
Record Dates: First submitted 2025-07-09; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Visual impairment; New method for amblyopia screening; Pediatric amblyopia screening; Eye Tracking system
MeSH Terms: conditions — Amblyopia; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amblyopic patient: Patient aged between 3 and 7 years, with amblyopia diagnosed by standard reference screening within the three months preceding the signing of the informed consent form.
  Interventions: Diagnostic Test: Standard screening procedure for amblyopia; Diagnostic Test: New amblyopia screening method using a virtual reality headset.
- Non Amblyopic patient: Patient aged between 3 and 7 years, non-amblyopic, who underwent routine screening confirming the absence of amblyopia or any other ocular condition that could lead to amblyopia, within the three months prior to signing the informed consent form.
  Interventions: Diagnostic Test: Standard screening procedure for amblyopia; Diagnostic Test: New amblyopia screening method using a virtual reality headset.

INTERVENTIONS:
Diagnostic Test: Standard screening procedure for amblyopia — The standard examination for amblyopia screening consists of three steps:
  A monocular visual acuity assessment using optotypes from the LEA scale, presented from the simplest to the most complex in front of each eye via an alternating occlusion mask.
  A cover/uncover test, during which the child is required to fixate on an image A Lang I stereopsis test performed under binocular vision.
Diagnostic Test: New amblyopia screening method using a virtual reality headset. — The examination with the virtual reality headset consists of three main steps: A monocular visual acuity assessment using optotypes from the LEA scale, presented from the simplest to the most complex in front of each eye via an alternating occlusion mask. The eye-tracking system analyzes fixation and the visual response of the stimulated eye. A cover/uncover test, during which the child is required to fixate on an image projected inside the headset. Eye movements are tracked to detect any deviations or abnormalities in ocular coordination. A Lang I stereopsis test performed under binocular vision, in which the child must identify three-dimensional images hidden within a virtual board. The eye-tracking system detects fixation on the images and allows evaluation of depth perception

SUMMARY:
Amblyopia, characterized by reduced visual acuity, develops in childhood due to insufficient sensory stimulation of the affected eye. It is the leading cause of low vision and loss of stereoscopic vision in both children and adults. Currently, 99 million people worldwide are affected, with recent projections indicating 222 million by 2040. Amblyopia can result from anisometropia (70%), strabismus (30%), or the presence of an ocular pathology (1%). Early management of these conditions (before the age of 7) can prevent the onset of amblyopia. Therefore, screening for these conditions is a major public health challenge to reduce the prevalence and associated costs of visual impairment.

The French-speaking Association of Strabology and Pediatric Ophthalmology (AFSOP) recommends systematic amblyopia screening for 3-year-old children. This screening involves measuring monocular visual acuity in both eyes (LEA chart at 3 meters), checking for strabismus (cover/uncover test), and performing a stereoscopic vision test (e.g., Lang I test).

Amblyopia is currently underdiagnosed for two main reasons: 1) it is often asymptomatic (75% of cases) and therefore cannot be detected without systematic screening; and 2) there is significant difficulty in accessing medical care in certain regions, and thus access to professionals capable of performing this screening (doctors, orthoptists). The difficulty in accessing healthcare professionals capable of screening for amblyopia in children aged 3 to 7 has already been raised.

We believe it would be beneficial to have an alternative screening method that is equivalent to the AFSOP-recommended method and accessible in areas with limited healthcare professionals. An eye-tracking system implemented in a virtual reality (VR) headset has recently been developed for monitoring eye movements. This system has shown effectiveness in rehabilitating visual field impairments in patients with traumatic brain injury. The system allows for remote monitoring of rehabilitation sessions, and data can be downloaded and viewed remotely via Wi-Fi.

The main objective of this study will be to estimate the sensitivity of the new VR-based eye-tracking screening method amblyopia screening method using an eye-tracking system implemented in a virtual reality headset compared to standard screening in children aged 3 to 7 years.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 3 to 7 years at the time of consent signing.
* Patients followed in the Ophthalmology Department of Strasbourg University Hospital (CHU Strasbourg).
* Holders of parental authority must be affiliated with or beneficiaries of the health insurance system.
* Holders of parental authority must be capable of understanding the objectives and risks related to the research, and able to provide dated and signed informed consent.
* Amblyopic patients must have amblyopia diagnosed by the reference screening method.
* Non-amblyopic patients must have undergone routine screening confirming the absence of amblyopia or any other ocular condition that could lead to amblyopia.
* Screening must be performed in the Ophthalmology Department of CHU Strasbourg, unless a prior screening has been performed according to established guidelines and fully documented in a report by the patient's ophthalmologist (detailed results of the three standard screening tests).
* The screening examination must have been performed within the three months prior to the signing of the informed consent form.

Exclusion criteria:

* Amblyopic children currently undergoing treatment or having previously received treatment for amblyopia (optical correction, strabismus surgery, occlusion therapy, orthoptic rehabilitation).
* Children presenting conditions or states that may cause side effects related to the use of the virtual reality headset (epilepsy, neurological or developmental disorders, autism spectrum disorders, dizziness, nausea, claustrophobia, etc.).
* Inability to provide informed information to the patient or holders of parental authority (emergency situations, difficulties in patient comprehension, etc.).

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3 to 7 years, including both amblyopic and non-amblyopic patients. All participants are recruited from the Ophthalmology Department of Strasbourg University Hospital (CHU Strasbourg) or referred by their ophthalmologists.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of a new amblyopia screening method compared to standard screening | At enrollment.
  Sensitivity of a new amblyopia screening method using an eye-tracking system implemented in a virtual reality headset, compared to standard screening, in children aged 3 to 7 years.
  Sensitivity = (true positives) / (false negatives + true positives)

SECONDARY OUTCOMES:
Specificity of the eye-tracking system compared to standard screening | At enrollment.
  Specificity of the eye-tracking system implemented in a virtual reality headset, compared to standard screening in children aged 3 to 7 years.
  Specificity = (true negatives) / (false positives + true negatives)
Sensitivity and specificity of the eye-tracking system compared to the same tests performed during standard screening | At enrollment.
  These are respectively:
  Monocular visual acuity of both eyes measured using the LEA symbol scale at 3 meters, presented via the virtual reality interface.
  Presence or absence of a refixation movement during the cover/uncover test for strabismus screening.
  Presence or absence of stereoscopic vision anomalies evaluated by projecting a Lang I test under binocular vision within the virtual reality headset.
Cover/uncover test for strabismus screening : angle of deviation | At enrollment.
  The angle of deviation of movement of each eye (refixation movement) will be recorded using a cover/uncover test combined with monocular stimulation
Proportion of adverse events recorded during the diagnostic process | Day of the diagnostic examination (Day 1)
  The proportion of adverse events will be recorded by the investigator accompanying the child during the examination with the virtual reality system across all study groups. In particular, adverse events related to the use of the virtual reality headset will be documented (nausea, discomfort, photophobia, seizure).
Proportion of patients unable to complete the scheduled examination using the virtual reality headset | Day of the diagnostic examination (Day 1)
  The proportion of patients unable to complete the scheduled examination using the virtual reality headset for any reason (including refusal to wear the headset, anxiety, or other factors) will be documented. This will include the number of patients for whom the examination could not be performed due to these reasons.
Cover/uncover test for strabismus screening : direction | At enrollment
  The direction of movement of each eye will be recorded using a cover/uncover test combined with monocular stimulation
Cover/uncover test for strabismus screening : velocity | At enrollment
  The velocity of movement of each eye (refixation movement) will be recorded using a cover/uncover test combined with monocular stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Misawa M, Bajin IY, Zhang B, Daibert-Nido M, Tchao D, Garcia-Giler E, Cheung K, Appel L, Nasir P, Reginald A, Tabori U, Bartels U, Ramaswamy V, Markowitz SN, Bouffet E, Reber M. A telerehabilitation program to improve visual perception in children and adolescents with hemianopia consecutive to a brain tumor: a single-arm feasibility and proof-of-concept trial. EClinicalMedicine. 2024 Nov 29;78:102955. doi: 10.1016/j.eclinm.2024.102955. eCollection 2024 Dec. PMID 39687429
- [Background] Daibert-Nido M, Pyatova Y, Cheung K, Nayomi C, Markowitz SN, Bouffet E, Reber M. Case Report: Visual Rehabilitation in Hemianopia Patients. Home-Based Visual Rehabilitation in Patients With Hemianopia Consecutive to Brain Tumor Treatment: Feasibility and Potential Effectiveness. Front Neurol. 2021 Jul 21;12:680211. doi: 10.3389/fneur.2021.680211. eCollection 2021. PMID 34354660
- [Background] Bois C, Milcent K, Dufourg M, Charles M. Bilan de santé des enfants de 3-4 ans en école maternelle par la Protection Maternelle Infantile en 2014-2016 : disparités départementales des pratiques. Bulletin Epidémiologique Hebdomadaire. Janvier 2020
- [Background] Lequeux L, Thouvenin D, Couret C, Audren F, Costet C, Dureau P, Leruez S, Defoordt-Dhellemmes S, Daien V, Espinasse Berrod MA, Arsene S, Lebranchu P, Denis D, Bui-Quoc E, Speeg-Schatz C. [Vision screening for children: Recommended practices from AFSOP]. J Fr Ophtalmol. 2021 Feb;44(2):244-251. doi: 10.1016/j.jfo.2020.07.005. Epub 2020 Dec 30. French. PMID 33388188
- [Background] Kaur S, Sharda S, Aggarwal H, Dadeya S. Comprehensive review of amblyopia: Types and management. Indian J Ophthalmol. 2023 Jul;71(7):2677-2686. doi: 10.4103/IJO.IJO_338_23. PMID 37417105
- [Background] Fu Z, Hong H, Su Z, Lou B, Pan CW, Liu H. Global prevalence of amblyopia and disease burden projections through 2040: a systematic review and meta-analysis. Br J Ophthalmol. 2020 Aug;104(8):1164-1170. doi: 10.1136/bjophthalmol-2019-314759. Epub 2019 Nov 8. PMID 31704700